CLINICAL TRIAL: NCT05963685
Title: Impact of a Standardized Alarming System on Treatment Times and Workflow in Stroke Patients With Interhospital Transfer for Thrombectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Munich Municipal Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: MT-ALARM
Record Dates: First submitted 2023-07-19; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Acute Ischemic Stroke
Keywords: mechanical thrombectomy, telestroke, drip and ship, interhospital transfer, communication
MeSH Terms: conditions — Ischemic Stroke; Communication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- pre implementation period: stroke patients transferred within the 6 months before introduction of the alarming system
- implementation period: stroke patients transferred within the 6 months after introduction of the alarming system
  Interventions: Other: standardized MT alarming system
- post implementation period: stroke patients transferred within the 6-12 months after introduction of the alarming system
  Interventions: Other: standardized MT alarming system

INTERVENTIONS:
Other: standardized MT alarming system — Standardized alarming system via telephone loop in the primary thrombectomy centre triggered immediately after decision to mechanical thrombectomy in stroke patients admitted in primary stroke centers
  Groups: implementation period; post implementation period

SUMMARY:
The aim of this study is to evaluate the impact of a standardized alarming system on treatment times and workflow in stroke patients with interhospital transfer for mechanical thrombectomy (MT). The main questions it aims to answer are:

* Is the implementation of a standardized alarming system associated with shorter transfer and treatment times?
* Is the implementation of a standardized alarming system associated with a better adherence on existing standard operating procedures for interhospital transfer? We will analyze data from our existing thrombectomy registry comparing time periods before and after introduction of the MT alarming system.

ELIGIBILITY:
Inclusion Criteria:

* age >= 18 years
* diagnosis of acute ischemic stroke
* indication for mechanical thrombectomy
* admission to one of 7 participating primary stroke centers within in the catchment area of the referral center

Exclusion Criteria:

* unclear indication for mechanical thrombectomy (patients admitted for perfusion imaging before decision for or against a MT)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute ischemic stroke patients admitted to one of 7 nonurban primary stroke centers with subsequent interhospital transfer to a referral center for mechanical thrombectomy in Southeast Bavaria, Germany.
Sampling Method: Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2022-09-16 (Actual); Primary Completion 2024-03-15 (Estimated); Study Completion 2024-03-15 (Estimated)

PRIMARY OUTCOMES:
decision-to-groin time | 24 hours
  time from decision for MT (while patient still in the primary stroke center) to groin puncture (start of mechanical thrombectomy procedure in the primary thrombectomy center)

SECONDARY OUTCOMES:
decision-to-departure time | 24 hours
  time from decision for MT to departure of the patient from primary stroke center (to the primary thrombectomy center)
decision-to-arrival time | 24 hours
  time from decision for MT to arrival of the patient at the primary thrombectomy center
arrival-to-groin time | 24 hours
  time from arrival of the patient at the primary thrombectomy center to groin puncture (start of mechanical thrombectomy procedure)
rate of refusal of transfer requests due to lack of capacity | 24 hours
  rate of patients that had to be transferred to a secondary thrombectomy center instead of the primary thrombectomy centre due to lack of capacity in the referral clinic
decision-to-transfer request time | 24 hours
  Time from decision for MT to request of emergency medical service for interhospital transfer
Periprocedural complications | 24 hours
  rate of periprocedural complications during MT
Successful outcome of MT (mTICI > 2b) | 24 hours
  rate of successfully performed MT (mTICI > 2b) of all patients with attempted MT
groin-to-recanalization time | 24 hours
  Time from groin puncture to successful recanalization
Adverse events within 7 days | 7 days
  Adverse events within the first 7 days after transfer to referral center

CONTACTS AND LOCATIONS:
Locations (1):
- Munich Municipal Hospital, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No
No plan to make IPD available to other researchers.